CLINICAL TRIAL: NCT00654576
Title: Effectiveness of Antipsychotic Combination With Psychosocial Intervention on Outcome of Patients With Schizophrenia:One-Year Follow up.
Brief Title: Effectiveness of Antipsychotic Combination With Psychosocial Intervention on Outcome of Patients With Schizophrenia
Acronym: ACPIOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Central South University (Other)
Collaborators: Shanghai Mental Health Center (Other); Sichuan University (Other); Capital Medical University (Other); Nanjing Medical University (Other); Jiangxi Mental Hospital (Unknown); Hunan Mental Hospital (Other); Guangzhou Mental Hospital (Other); Chongqing Metal Institute (Unknown); Henan Mental Hospital (Unknown)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2004BA720A22
Record Dates: First submitted 2008-04-03; First posted 2008-04-08 (Estimated); Last update posted 2008-04-08 (Estimated); Status verified 2008-04

CONDITIONS: Schizophrenia
Keywords: schizophrenia; antipsychotic; outcome; psychosocial intervention
MeSH Terms: conditions — Schizophrenia | interventions — Chlorpromazine; Sulpiride; Clozapine; Olanzapine; Risperidone; Quetiapine Fumarate; Psychosocial Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): the comparator arm will only receive one of the seven antipsychotic
  Interventions: Drug: Chlorpromazine, Sulpiride, Clozapine, Olanzapine, Risperidone, Quetiapine, Aripitrazole
- 2 (Experimental): the experimental group will receive one of the seven study drugs combination with psychosocial intervention
  Interventions: Behavioral: psychosocial intervention

INTERVENTIONS:
Drug: Chlorpromazine, Sulpiride, Clozapine, Olanzapine, Risperidone, Quetiapine, Aripitrazole — patient will receive one of the seven study drugs (Chlorpromazine, Sulpiride, Clozapine, Olanzapine, Risperidone, Quetiapine, Aripitrazole) as the maintain treatment. the dose is flexible, is based on the study doctor's judgment.
  Arms: 1
Behavioral: psychosocial intervention — the psychosocial interventions include psychoeducaiton, family intervention, skill training, and cognitive-behavioral therapy.
  Arms: 2

SUMMARY:
Antipsychotic alone is limit to improve the overall outcome of schizophrenia and has a high discontinue rate.To solve these problems, we provide practical and available psychosocial intervention. We hypothesize that there will be significant difference in the overall effectiveness between antipsychotic and antipsychotic combination with psychosocial intervention.

DETAILED DESCRIPTION:
The study is designed as a national, multicenter, randomized, naturalistic trial, with research assessors intended to be blind to the intervention status.

We plan to recruit 1400 patients at 10 china sites and randomly assign them to two group. the control group only receive antipsychotic and the study group receive antipsychotic combination with psychosocial intervention. The course is 12 months. Patients use one of the seven study drugs (chlorpromazine, sulpiride, clozapine, olanzapine, risperidone, quetiapine, and aripitrazole)to the maintain treatment. The psychosocial intervention include psychoeducation, family intervention, skills training, and cognitive-behavioral therapy. The primary aim is to delineate differences in the overall effectiveness of the two treatment model.The assessments include the outcome of symptomatology，neurobiology，social psychology，medical economics.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients were 16 to 50 years of age;
* had received a diagnosed of schizophrenia in accordance with criteria set out in the Diagnostic and Statistical Manual of Mental Disorders-fourth edition (DSM-IV);
* were confirmed to be clinically stable by the investigator (the total score ≤60 on the Positive and Negative Syndrome Scale [PANSS] or a decrease of fifty percent from acute period in the total score on PANSS)
* and taken maintenance treatment with any one of the following seven oral antipsychotics:

  * chlorpromazine
  * sulpiride clozapine
  * risperidone
  * olanzapine
  * quetiapine
  * aripiprazole

Exclusion Criteria:

* Patients were excluded if they had received a diagnosis of schizoaffective disorder, mental retardation, or other cognitive disorders;
* had a history of serious adverse reactions to the proposed treatment;
* were pregnant or breastfeeding; or had a serious and unstable medical condition.
* Patients were excluded if they were unable to provide informed consent

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1400 (Estimated)
Dates: Start 2005-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
the time to discontinued treatment and the rate of relapse/rehospitalization

SECONDARY OUTCOMES:
clinical psychopathology, side effect, compliance, social function, neurocognitive function, quality of life, family/career burden, cost analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Mental Health of The Second Xiangya Hospital, Central South University, Changsha, Hunan, China

REFERENCES:
- [Derived] Zhang Z, Zhai J, Wei Q, Qi J, Guo X, Zhao J. Cost-effectiveness analysis of psychosocial intervention for early stage schizophrenia in China: a randomized, one-year study. BMC Psychiatry. 2014 Jul 26;14:212. doi: 10.1186/s12888-014-0212-0. PMID 25064681
- [Derived] Guo X, Fang M, Zhai J, Wang B, Wang C, Hu B, Sun X, Lv L, Lu Z, Ma C, Guo T, Xie S, Twamley EW, Jin H, Zhao J. Effectiveness of maintenance treatments with atypical and typical antipsychotics in stable schizophrenia with early stage: 1-year naturalistic study. Psychopharmacology (Berl). 2011 Aug;216(4):475-84. doi: 10.1007/s00213-011-2242-3. Epub 2011 Mar 3. PMID 21369751
- [Derived] Guo X, Zhai J, Liu Z, Fang M, Wang B, Wang C, Hu B, Sun X, Lv L, Lu Z, Ma C, He X, Guo T, Xie S, Wu R, Xue Z, Chen J, Twamley EW, Jin H, Zhao J. Effect of antipsychotic medication alone vs combined with psychosocial intervention on outcomes of early-stage schizophrenia: A randomized, 1-year study. Arch Gen Psychiatry. 2010 Sep;67(9):895-904. doi: 10.1001/archgenpsychiatry.2010.105. PMID 20819983